CLINICAL TRIAL: NCT02834442
Title: A Randomised, Double Blind, Placebo Controlled Phase I Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of MT-7117 in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of MT-7117 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-7117-E01
Record Dates: First submitted 2016-07-06; First posted 2016-07-15 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Healthy

ARMS (2):
- Single ascending dose, MT-7117 or Placebo (Experimental)
  Interventions: Drug: MT-7117; Drug: Placebo
- Multiple ascending dose, MT-7117 or Placebo (Experimental)
  Interventions: Drug: MT-7117; Drug: Placebo

INTERVENTIONS:
Drug: MT-7117
Drug: Placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of MT-7117 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free from clinically significant illness or disease
* Male or female subjects aged 18 to 55 years or elderly male subjects aged ≥65
* A body weight of ≥60 kg for males and ≥50 kg for females, and a body mass index ranging from 18 to 30 kg/m2

Exclusion Criteria:

* Participated in more than three clinical studies involving administration of an IMP in the previous year, or any study within 12 weeks
* Clinically significant endocrine, thyroid, hepatic, respiratory, gastro intestinal, renal, cardiovascular or skin disease, or history of any significant psychiatric/psychotic illness disorder
* Clinically relevant abnormal medical history, physical findings or laboratory values

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as measured by number of participants with adverse events | up to Day56
Safety and Tolerability as measured by vital signs | up to Day56
Safety and Tolerability as measured by physical examination | up to Day56
Safety and Tolerability as measured by ECG | up to Day21
Safety and Tolerability as measured by laboratory safety assessments | up to Day21

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 96 hours post dose
Area under the plasma concentration-time curve (AUC) | 96 hours post dose
Time to maximum plasma concentration (Tmax) | 96 hours post dose
Apparent elimination half-life in plasma | 96 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational center, United Kingdom, United Kingdom

REFERENCES:
- [Derived] Ogasawara A, Ide R, Inoue S, Tsuda M, Teng R. Assessment of Potential Drug-Drug Interactions for Novel Oral Melanocortin-1 Receptor Agonist Dersimelagon. Pharmacol Res Perspect. 2025 Feb;13(1):e70069. doi: 10.1002/prp2.70069. PMID 39887900
- [Derived] Ogasawara A, Ogawa K, Ide R, Ikenaga Y, Fukunaga C, Nakayama S, Tsuda M. Results from a first-in-human study of dersimelagon, an investigational oral selective MC1R agonist. Eur J Clin Pharmacol. 2023 Jun;79(6):801-813. doi: 10.1007/s00228-023-03476-6. Epub 2023 Apr 15. PMID 37060458